CLINICAL TRIAL: NCT03145961
Title: c-TRAK TN: A Randomised Trial Utilising ctDNA Mutation Tracking to Detect Minimal Residual Disease and Trigger Intervention in Patients With Moderate and High Risk Early Stage Triple Negative Breast Cancer
Brief Title: A Trial Using ctDNA Blood Tests to Detect Cancer Cells After Standard Treatment to Trigger Additional Treatment in Early Stage Triple Negative Breast Cancer Patients
Acronym: c-TRAK-TN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: National Institute for Health Research Biomedical Research Centre at the Royal Marsden / Institute of Cancer Research UK (Unknown); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICR-CTSU/2016/10058; 2017-000508-92 (EudraCT Number)
Record Dates: First submitted 2017-04-28; First posted 2017-05-09 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Triple Negative Breast Cancer
Keywords: Breast cancer early stage; circulating tumour DNA; pembrolizumab; targeted therapy; randomised clinical trial; phase II; mutation screening; intermediate endpoint
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: atients will undergo blinded serial ctDNA screening every 3 months from the point of registration and completion of primary treatment for their triple negative breast cancer. If a ctDNA positive result occurs on or before their 12 month ctDNA screening assessment the patient will be randomised by the ICR-CTSU in a 2:1 ratio to the pembrolizumab treatment arm or observation arm. The patient and their treating team will only be informed of the randomisation if they are allocated to the treatment arm.
  For patients allocated to the observation group, the treating team and patient will not be informed that randomisation has taken place in order to remain blinded to the positive ctDNA result. Such patients will continue to have blood samples collected for ctDNA analysis every 3 months up to 2 years from starting ctDNA screening.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Observation (No Intervention): Patient will have blood samples collected for ctDNA analysis every 3 months for up to 2 years from starting ctDNA screening.
- Pembrolizumab Treatment (Experimental): Patients will be given pembrolizumab every 3 weeks for up to a maximum of 12 months, with blood samples collected prior to each cycle for continued ctDNA analysis. Following treatment discontinuation, blood samples will be collected for ctDNA analysis every 3 months for a further 12 months.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — 200mg intravenous infusion
  Other Names: Keytruda
  Arms: Pembrolizumab Treatment

SUMMARY:
c-TRAK TN is a multi-centre phase II study, consisting of a circulating tumour DNA (ctDNA) surveillance component and a therapeutic component. c-TRAK TN aims to assess whether ctDNA surveillance can be used to detect residual disease following patients standard primary treatment for triple negative breast cancer, and will assess the safety and activity of the investigational medicinal product pembrolizumab.

DETAILED DESCRIPTION:
During the randomised component of the trial (prior to implementation of protocol v6.0 on 16 Sept 2020), patients would undergo serial ctDNA surveillance every 3 months from the point of registration and completion of primary treatment for their triple negative breast cancer. ctDNA surveillance was blinded and the detection of a ctDNA positive result on or before the 12 month ctDNA surveillance assessment triggered randomisation to treatment with pembrolizumab or observation (on a 2:1 ratio). The patient and their treating team were only informed of the randomisation if allocated treatment.

Patients without a positive ctDNA result within 12 months of starting ctDNA surveillance, continued to have blinded ctDNA surveillance every 3 months up to 2 years total.

Following the implementation of protocol v6.0 (16 Sept 2020), patients were asked to transfer to the non-randomised component of the trial, all patients who were previously randomised to observation and remain in active ctDNA surveillance would transition to the non-randomised component of the trial following re-consent, and allocated pembrolizumab at the next positive ctDNA result.

All patients will be followed up every 6 months until disease recurrence, specific withdrawal of consent for follow up, or until sponsor advises no further follow up is required.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form for Registration.
2. Male or female patients ages 16 years or older.
3. ECOG performance status 0, 1 or 2.
4. Histologically proven primary triple negative breast cancer as defined as oestrogen receptor (ER) negative, progesterone receptor (PgR) negative (if available, otherwise PgR unknown), (as defined by Allred score 0/8 or 2/8 or stain in <1% of cancer cells) and HER2 negative (immunohistochemistry 0/1+ or negative by in situ hybridization) as determined by local laboratory.
5. Availability of tissue from two archival tumour tissue samples (either from diagnostic biopsy and/or primary surgery). If only one tumour sample is available, the site should inform the ICR-CTSU who will discuss eligibility with the Chief Investigator (or designated TMG member). Patients who have tumours previously sequenced outside the c-TRAK TN trial must provide one archival tumour tissue sample and the report that confirms the mutations detected.
6. Patients with moderate or high risk early stage triple negative breast cancer according to the following risk of relapse criteria:

   Neoadjuvant chemotherapy (no adjuvant chemotherapy planned) High risk criteria - Residual microscopic or macroscopic invasive cancer in the axillary nodes after chemotherapy Moderate risk criteria - Residual invasive cancer in the breast, and axillary lymph node negative after chemotherapy Adjuvant chemotherapy High risk criteria - Tumour size >50mm and node positive OR ≥4 nodes positive regardless of primary tumour size.

   Moderate risk criteria - Tumour size >20mm AND/OR involved axillary macroscopic lymph node.

   Both neoadjuvant and adjuvant chemotherapy Patients who have received both neoadjuvant chemotherapy and further adjuvant chemotherapy must fulfil only the adjuvant chemotherapy risk criteria to be eligible. They can fulfil the criteria on either clinical staging prior to neoadjuvant chemotherapy or pathological staging at surgery.
7. Patients must be registered according to the following criteria for timing of registration:

   Neoadjuvant chemotherapy (no adjuvant chemotherapy planned):

   Patients must be registered within 6 weeks of surgery. Patients may be registered before or during radiotherapy and should be registered as early as possible.

   Adjuvant chemotherapy (no neoadjuvant chemotherapy received):

   Patients must be registered before, or on the day of, the 3rd cycle of adjuvant chemotherapy and should be registered as early as possible.

   Both neoadjuvant and adjuvant chemotherapy Patients must be registered within 6 weeks of surgery. Patients may be registered before or during radiotherapy. Patients must register before starting capecitabine.
8. Consent to provide research blood samples.
9. Patients with bilateral tumours can be included if both are triple negative and if two archival tissues samples can be provided per tumour.
10. Patients must have had surgery achieving clear margins (as per local guidelines).
11. Female and male patients of reproductive potential must be willing to use an adequate method of contraception for the first year of the trial and, if allocated to pembrolizumab, for the duration of treatment through to 120 days after the last dose of pembrolizumab (see appendix 2). Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient.
12. Patients must be willing to have frequent blood tests (every 3 months for 2 years in ctDNA surveillance and 3 weekly if subsequently allocated pembrolizumab) and receive a 12 month course of pembrolizumab on ctDNA detection.
13. No evidence of distant metastatic disease or local recurrence on staging scans conducted at any time since initial diagnosis.

NB: Additional eligibility criteria apply to confirm eligibility to commence pembrolizumab treatment following randomisation.

Exclusion Criteria:

1. Any concurrent or planned treatment for the current diagnosis of breast cancer other than surgery, loco regional adjuvant radiotherapy, standard neoadjuvant or adjuvant chemotherapy, or a bisphosphonate/denosumab.
2. Prior treatment with a PDL1, PD1, or other immunomodulatory therapy.
3. Prior diagnosis of cancer (including prior diagnosis of breast cancer) in the previous 5 years, other than for basal cell carcinoma of the skin or cervical carcinoma in situ.
4. Patients previously entered into a therapeutic trial during or after neoadjuvant chemotherapy where experimental therapy is continued post-surgery (see protocol section 15).
5. Treatment with an unlicensed or investigational product within 4 weeks of trial entry.
6. Active autoimmune disease requiring systemic therapy in the last two years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of such systemic treatment.
7. Diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of pembrolizumab.
8. Known history of active Tuberculosis Bacillus (TB).
9. Known history of Human Immunodeficiency Virus (HIV).
10. Known active Hepatitis B or Hepatitis C.
11. Known history of, or any evidence of active, non-infectious pneumonitis.
12. Active infection requiring systemic therapy.
13. Previous solid organ or allogenic stem cell transplantation.
14. Females who are pregnant or breastfeeding.
15. Presence of any systemic illness incompatible with participation in the clinical trial or inability to provide written informed consent.
16. A pathological complete response (pCR) to neoadjuvant chemotherapy

NB. Additional exclusion criteria apply to confirm eligibility to commence pembrolizumab treatment following randomisation.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Positive ctDNA detection by 12 months | 12 months
  The proportion of patients with ctDNA positivity by 12 months as assessed by the blood sample taken at that timepoint
Positive ctDNA detection by 24 months | 24 months
  The proportion of patients with ctDNA positivity by 24 months as assessed by the blood sample taken at that timepoint
Absence of detectable ctDNA or disease recurrence 6 months (24 weeks) after commencing pembrolizumab | 6 months (24 weeks) after commencing pembrolizumab
  The proportion of patients without either detectable ctDNA or disease recurrence 6 months (24 weeks) after starting pembrolizumab

SECONDARY OUTCOMES:
Time to ctDNA detection | Baseline to first ctDNA positivity (up to a maximum of 12 months after starting ctDNA surveillance)
  The time from entry into ctDNA surveillance to first positive ctDNA detection
Detection of overt metastatic disease at time of first ctDNA detection in patients allocated to pembrolizumab | Baseline to first ctDNA positivity (up to a maximum of 12 months after starting ctDNA surveillance)
  Proportion of patients with metastatic disease at the same time point as first positive ctDNA detection
Lead time between ctDNA detection and disease recurrence in the pembrolizumab treatment and observation groups | From date of randomisation to recurrence detection, expected to occur up to 5 years
  The time between randomisation to the therapeutic aspect of the trial (either to pembrolizumab treatment or observation group) and first confirmed detection of recurrent disease.
Absence of detectable ctDNA or disease recurrence after 6 months in the observation group | 6 months after randomisation
  Proportion of patients without detectable ctDNA or disease recurrence 6 months after randomisation to observation group
Safety and tolerability of pembrolizumab assessed using NCI CTCAE v4.0, and the proportion of patients reporting dose reductions or delays. | Throughout pembrolizumab treatment, up to 12 months of treatment
  Adverse events assessed throughout treatment period, using the NCI CTCAE v4.0. Proportion of patients reporting a dose reduction or delay will be presented.
Commencement of treatment in patients randomised to receive pembrolizumab | At point of commencement or non-commencement of treatment, up to 8 weeks following randomisation
  Proportion of patients randomised to receive pembrolizumab who start the therapy.

OTHER OUTCOMES:
Descriptive differences in time between ctDNA detection and disease recurrence, and disease free survival, between patients in the pembrolizumab and the observation groups | Time between first ctDNA detection and documented recurrence or disease free survival event, whichever comes first, expected to occur up to 5 years
  Time from first positive ctDNA detection to disease recurrence or disease-free survival event.
To explore predictors of sustained ctDNA clearance on pembrolizumab. | 6-12 months after commencing pembrolizumab
  The relationship between sustained clearance of ctDNA on pembrolizumab and biological markers will be summarised and investigated using logistic regression.
To explore potential predictors of relapse and ctDNA detection, and alternative definitions of ctDNA clearance | Baseline to point of disease recurrence, expected to occur up to 5 years
  Relationship between lead time and clinical/biological factors will be assessed using standard statistical techniques for time to event data.
Association between ctDNA clearance and time to recurrence in pembrolizumab group | Time of ctDNA clearance to time of recurrence, expected to occur up to 5 years
  Relationship between ctDNA clearance and time to recurrence in the pembrolizumab group will be assessed using standard statistical techniques for time to event data.

CONTACTS AND LOCATIONS:
Overall Officials: Nick Turner, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (17):
- United Kingdom (17):
  - Royal Marsden Hospital, Chelsea, Chelsea, London
  - Royal Marsden Hospital, Sutton, Sutton, Surrey
  - Royal Bournemouth Hospital, Bournemouth
  - Velindre Cancer Centre, Cardiff
  - Western General Hospital, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Guy's Hospital, London
  - Charing Cross Hospital, London
  - St Bartholomew's Hospital, London
  - University College London Hopitals, London
  - Maidstone Hospital, Maidstone
  - The Christie NHS Foundation Trust, Manchester
  - Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Churchill Hospital, Oxford
  - Weston Park Hospital, Sheffield
  - Royal Cornwall Hospital, Truro

IPD SHARING:
Plan to Share IPD: Undecided
Formal requests for data sharing will be considered in line with ICR-CTSU procedure with due regard given to funder and sponsor guidelines. Requests are via a standard pro forma describing the nature of the proposed research and extent of data requirements. Data recipients are required to sign a data release form which describes the conditions for release and requirements for data transfer, storage, archiving, publication and Intellectual Property.

REFERENCES:
- [Derived] Turner NC, Swift C, Jenkins B, Kilburn L, Coakley M, Beaney M, Fox L, Goddard K, Garcia-Murillas I, Proszek P, Hall P, Harper-Wynne C, Hickish T, Kernaghan S, Macpherson IR, Okines AFC, Palmieri C, Perry S, Randle K, Snowdon C, Stobart H, Wardley AM, Wheatley D, Waters S, Winter MC, Hubank M, Allen SD, Bliss JM; c-TRAK TN investigators. Results of the c-TRAK TN trial: a clinical trial utilising ctDNA mutation tracking to detect molecular residual disease and trigger intervention in patients with moderate- and high-risk early-stage triple-negative breast cancer. Ann Oncol. 2023 Feb;34(2):200-211. doi: 10.1016/j.annonc.2022.11.005. Epub 2022 Nov 22. PMID 36423745